CLINICAL TRIAL: NCT04389866
Title: Jowl Improvement With Injectable Fillers: Jawline Injections Alone vs Jawline and Cheek Injections
Brief Title: Jowl Improvement With Injectable Fillers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Advanced Dermatology (Other)
Collaborators: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10001 Jowl Voluma
Record Dates: First submitted 2020-04-29; First posted 2020-05-15 (Actual); Results first posted 2024-02-15 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-01

CONDITIONS: Jowls
Keywords: Jowls; Lower Face Laxity; Filler; JUVÉDERM VOLUMA™ XC.; Melolabial Folds; Wrinkles

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Both Jawline and Lateral (Zygomatic) Cheek Area Injections (Experimental): JUVÉDERM VOLUMA™ XC 1-3 syringes (each syringe is 1 cc) will be injected bilaterally into the lateral cheek (zygomatic) area plus JUVÉDERM VOLUMA™ XC 1-2 syringes (each syringe is 1 cc) will be injected into the lateral jawline and inferior cheek area (preauricular area) (the latter area will be added if necessary to achieve visual improvement in jowl attenuation). Total syringes used per person will have a range of 2-5)
  Interventions: Device: JUVÉDERM VOLUMA™ XC
- Jawline Injections (Experimental): JUVÉDERM VOLUMA™ XC 1-2 syringes (each syringe is 1 cc) will be injected bilaterally into the lateral jawline and inferior cheek area (preauricular area) (the latter area will be added if necessary to achieve visual improvement in jowl attenuation). Total syringes used per person will have a range of 1-2)
  Interventions: Device: JUVÉDERM VOLUMA™ XC

INTERVENTIONS:
Device: JUVÉDERM VOLUMA™ XC — Injectable gel
  Other Names: non-animal hyaluronic acid

SUMMARY:
This is a prospective clinical study to demonstrate a reduction in jowling and laxity of the jawline that can be achieved following facial volume enhancement using JUVÉDERM VOLUMA™ XC (0.3% w/w lidocaine). The secondary measure will be if this can be achieved with Jawline injection only, or if a superior result can be obtained with both cheek and jowl injection.

DETAILED DESCRIPTION:
This study is proposed to evaluate the best protocol for achieving improvement in the sagging jawline.

JUVÉDERM VOLUMA™ XC will be injected in each of 16 women with sagging of grades 1-3 using a published jawline evaluation scale.

Patients will be randomized into 1:1 into 2 groups:

Patient Group 1: JUVÉDERM VOLUMA™ XC 1-2 syringes (each syringe is 1 cc) will be injected bilaterally into the lateral jawline and inferior cheek area (preauricular area) (the latter area will be added if necessary to achieve visual improvement in jowl attenuation). Total syringes used per person will have a range of 1-2)

Patient Group 2: JUVÉDERM VOLUMA™ XC 1-3 syringes (each syringe is 1 cc) will be injected bilaterally into the lateral cheek (zygomatic) area plus JUVÉDERM VOLUMA™ XC 1-2 syringes (each syringe is 1 cc) will be injected into the lateral jawline and inferior cheek area (preauricular area) (the latter area will be added if necessary to achieve visual improvement in jowl attenuation). Total syringes used per person will have a range of 2-5)

High-resolution photographs from multiple angles will be taken in identical lighting and position with the VISIA CR (clinical research) and with the Fotofinder at baseline, 2 weeks, 4 weeks, 8 weeks, and 12 or 16 weeks. Additional real-time video telemedicine visits will take place at 6 months and 12 months. In addition, a 72-hour safety phone call will be completed with the subject after each injection session. All visit timing will be based on the last injection session. One blinded dermatologist and one unblinded dermatologist will rate the patient's severity of jowling based on the Jawline Rating Scale (JRS) (1) at the 4-week, 8-week, and either 12 or 16-week visits. The patient will also rate their jowling based on the JRS as well as their satisfaction with the procedure.

ELIGIBILITY:
Inclusion Criteria

1. Jowling grade 2-3 by the Lower Face Jawline at Rest Scale (1), by both MD evaluator and patient.
2. Female patients must not be pregnant or trying to get pregnant and must have negative pregnancy tests before treatment.
3. Non-pregnant females ages 35-75 in good general health.
4. A study participant must be able to give proper informed consent in writing and be willing to follow the treatment schedule and undertake to carry out all necessary precautions and instructions.
5. Able to participate in telemedicine video visits.
6. Able to understand the requirements of the study and willing and able to follow all study procedures and attend all study visits, and successfully complete the study.
7. Willing to refrain from any other cosmetic procedures on the face including surgery, thread lifting, botulinum toxin in the masseters, jawline, neck, lips or chin, chemical peels, lasers or energy-based devices meant to improve volume or laxity of the face, and additional injectable fillers from the first visit through 12 months after last injection session.

Exclusion Criteria

1. Pregnancy or nursing
2. Hyaluronic acid filler injections in the past 6 months in the lower face or unwilling to refrain from such injections other than in the study for the duration of the study.
3. Radiesse or Sculptra in the past 24 months in the lower face
4. Permanent fillers or injectable fat at any time in the past.
5. Facial surgery, tissue tightening, or laser treatments within the past 24 months in the lower face, or unwilling to refrain from having these treatments for the duration of the study.
6. History of keloid or scar formation
7. Unwillingness to refrain from excessive sun exposure or tanning beds during the healing process
8. Taking any medications or supplements that will increase the potential for bruising, or discontinuation of same for 10 days prior to the procedure if medically allowed. These include but are not limited to aspirin of any dosage, any prescription blood thinner, vitamin E, and fish oil.
9. Any of the following significant medical problems: diabetes, obesity, autoimmune disease, cancer, inflammation at the site of injection, current infection any place on the body, dental work in the prior 2 weeks or scheduled for the post-treatment 2-week period, dementia, facial nerve abnormalities, history of blood clots, Bell's Palsy or any neurological condition affecting the facial muscles or nerves.
10. Prior tattoos, piercings, facial hair, or scars below and including the subnasal area that could interfere with visual assessment of the chin, jowls, jawline, and could promote bias in the evaluation of improvement or safety.
11. Known allergy or sensitivity to any components of the injection material, lidocaine, or hyaluronidase.
12. Current enrollment in any other investigational drug or device trial.
13. Any condition that the investigator believes might interfere with study results or put the subject at significant risk with participation.
14. Patients planning to undergo any dental procedure (other than prophylaxis and dental) fillings) during the study will be excluded in order to reduce risks related to seeding infection during injections.
15. Patients who have undergone mesotherapy or cosmetic treatment (laser, photomodulation, intense pulsed light, radiofrequency, dermabrasion, moderate or greater depth chemical peel, liposuction, lipolysis, or other ablative procedures) anywhere in the face or neck, or botulinum toxin treatment below the subnasal region (including injections to the masseter muscles) within 6 months before enrollment or was planning to undergo any of these procedures during the study.
16. Patients who experienced trauma to the chin and jaw area within 6 months before enrollment or had residual deficiencies, deformities, or scarring.
17. Patients with a history of anaphylaxis or allergy to lidocaine (or any amide-based anesthetics), hyaluronic acid products, or Streptococcal protein, or was planning to undergo desensitization therapy during the term of the study.
18. Patients who had porphyria, untreated epilepsy, or active autoimmune disease.
19. Patients who had current cutaneous or mucosal inflammatory or infectious processes (e.g., acne, herpes, gum disease), abscess, an unhealed wound, or a cancerous or precancerous lesion, below the subnasal (study device injection may have been delayed for participants with a history of recurrent oral herpes lesions who take prophylactic doses of antiviral/herpes medication for at least 2 days before study treatment administration)
20. Patients on a concurrent regimen of lidocaine or structurally-related local anesthetics (e.g., bupivacaine) or was on a concurrent regimen of drugs that reduce or inhibit hepatic metabolism (e.g., cimetidine, beta-blockers)
21. Patients on a regimen of anticoagulation therapy (e.g., warfarin, clopidogrel) or other prescription anticoagulation therapy.
22. Patients on a regimen of medications (e.g., aspirin or ibuprofen) or other substances known to increase coagulation time (e.g., herbal supplements with garlic or Gingko Biloba) within 10 days of undergoing study device injection (study device injection may have been delayed as necessary to accommodate this 10-day washout period)
23. Patients who received any investigational product within 30 days prior to study enrollment or were planning to participate in another investigation during the course of this study.
24. Patients who have begun using any new over-the-counter or prescription oral or topical, anti-wrinkle products below the subnasal area within 30 days before enrollment or was planning to begin using such products during the study (participants who had been on a regimen of such products for at least 30 days were eligible for the study if they intended to continue their regimen throughout the study).

Ages: 35 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2020-09-25 (Actual); Primary Completion 2022-10-05 (Actual); Study Completion 2022-10-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy Taub, MD, Principal Investigator — Advanced Dermatology
Locations (1):
- Advanced Dermatology, Lincolnshire, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited based on physician referral and review of clinic's electronic medical records at one clinical medical center between August 2020 and August 2021. The first participant was enrolled on September 25, 2020 and the last participant was enrolled in September 2021.
Pre-assignment Details: Photographs were obtained prior to randomization and treatment.
Groups:
- Jawline Injections: JUVÉDERM VOLUMA™ XC 1-2 syringes (each syringe is 1 cc) will be injected bilaterally into the lateral jawline and inferior cheek area (preauricular area) (the latter area will be added if necessary to achieve visual improvement in jowl attenuation). Total syringes used per person will have a range of 1-2) JUVÉDERM VOLUMA™ XC: Injectable gel
Period: Overall Study
Arm/Group | Jawline Injections | Both Jawline and Lateral (Zygomatic) Cheek Area Injections
Started | 8 | 8
Completed | 7 | 7 (Subject withdrew after screen.)
Not Completed | 1 | 1
Not completed — Patient with COVID-19 exposure concerns 03Dec2020 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Female subjects with jowls with severity grade 2-3 on the Merz Jawline Scale.
Groups:
- Total: Total of all reporting groups
Arm/Group | Jawline Injections | Both Jawline and Lateral (Zygomatic) Cheek Area Injections | Total
Number analyzed (Participants) | 7 | 7 | 14
Age, Continuous [Mean (Full Range); unit: years] | 53.65 [48.36 to 58.22] | 59.47 [46.076 to 63.277] | 56.92 [46.076 to 63.277]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 14
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White, non-hispanic | 6 | 7 | 13
  White, hispanic | 1 | 0 | 1
Moderate to Severe Jowl Severity [Mean (Standard Deviation); unit: Jawline Rating Scale units. Range 0 to 4] — Name of scale and what it measures:
  Merz Jawline Rating Scale which measures the degree of Jowl sagging.
  Scale range:
  0 = No sagging
  1. = Mild sagging
  2. = Moderate sagging
  3. = Severe sagging
  4. = Very Severe sagging
  Better outcome:
  Reduced sagging/lower number on scale
  Jawline Rating Scale units. Range 0 to 4 | 2.214 (.699) | 2.071 (.616) | 2.143 (.651)

OUTCOME MEASURES:

1. Primary Outcome: Blinded Physician Jawline Rating Scale (JRS) Assessment on Scale of 0 to 4 at Baseline Versus 4 Weeks After Last Injection.
Description: The primary outcome is a reduction of 1 or more points of the Jawline Rating Scale (JRS) Assessment (on a scale of 0 to 4) at baseline versus that at 4 weeks from the last injection (whether initial or touch-up) based on one blinded dermatologist rating. (A lower number will mean a better outcome) All subject data in respective groups were averaged into a single value at each time point.
  To clarify the Time Point "4 Weeks from last injection" it means 8 to 12 weeks after baseline as subjects were eligible for treatment 4 weeks after baseline and possible retreatment 8 weeks after baseline. The study wanted to capture results 4 weeks after last injection.
Time Frame: Baseline to 4 weeks after last injection.
Population: Intent to treat population (participants assigned to jawline injections versus both jawline and lateral (zygomatic) cheek area injections).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Jawline Injections | Both Jawline and Lateral (Zygomatic) Cheek Area Injections
Number analyzed (Participants) | 7 | 7
score on a scale
  Mean Jawline Rating Scores at baseline | 2.214 (.699) | 2.071 (.616)
  Mean Jawline Rating Scores at 4 weeks after last injection | 1.857 (0.864) | 1.857 (0.864)
  Reduction in Jawline rating score Baseline vs 4 Weeks after last injection | .357 (.864) | .214 (.864)
Statistical Analysis 1: Comparison: Jawline Injections; The null hypothesis for the 7 participants placed randomly 1:1 in the jawline injection arm was that there would be no statistically significant change in the blinded physician Jawline Rating Scale Assessment at baseline versus four weeks after last injection; Test type: Superiority; p = 0.018, t-test, 2 sided — The threshold for statistical significance was p = 0.05; The df = 13 for arm 1 (jawline injections) analysis of Jawline Rating Scale Assessments given by blinded physician; Mean Difference (Final Values) = -0.357, Standard Deviation 0.864 — Treatment Difference = 4 Weeks after last injection - Baseline
Statistical Analysis 2: Comparison: Both Jawline and Lateral (Zygomatic) Cheek Area Injections; The null hypothesis for the 7 participants placed randomly 1:1 in the jawline and lateral (zygomatic) cheek area injections arm was that there would be no statistically significant change in the blinded physician Jawline Rating Scale Assessment at baseline versus four weeks after last injection; Test type: Superiority; p = 0.082, t-test, 2 sided — The threshold for statistical significance was p = 0.05; The df = 13 for arm 2 (jawline and lateral zygomatic cheek area injections) analysis of Jawline Rating Scale Assessments given by blinded physician; Mean Difference (Final Values) = -0.214, Standard Deviation 0.864 — Treatment Difference = 4 Weeks after last injection - Baseline

2. Secondary Outcome: Unblinded Physician Jawline Rating Scale (JRS) Assessment on Scale of 0 to 4 at Baseline Versus 4 Weeks After Last Injection.
Description: One of the secondary outcomes is a reduction of 1 or more points of the Jawline Rating Scale (JRS) Assessment (on a scale of 0 to 4) at baseline versus that at 4 weeks from the last injection (whether initial or touch-up) based on one unblinded dermatologist rating. (A lower number will mean a better outcome).
  To clarify the Time Point "4 Weeks from last injection" it means 8 to 12 weeks after baseline as subjects were eligible for treatment 4 weeks after baseline and possible retreatment 8 weeks after baseline. The study wanted to capture results 4 weeks after last injection.
  Scale Range Description 0 = No sagging
  1. = Mild sagging
  2. = Moderate sagging
  3. = Severe sagging
  4. = Very Severe sagging
Time Frame: Baseline to 4 weeks after last injection.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Jawline Injections | Both Jawline and Lateral (Zygomatic) Cheek Area Injections
Number analyzed (Participants) | 7 | 7
score on a scale
  Mean Jawline Rating Scores at Baseline | 2.357 (0.497) | 2.357 (0.497)
  Mean Jawline Rating Scores at 4 weeks after last injection | 1.357 (0.497) | 1.643 (0.497)
  Mean Reduction in Jawline Rating Score Baseline vs 4 Weeks after last injection | 1.0 (0.497) | .714 (0.497)
Statistical Analysis 1: Comparison: Jawline Injections; The null hypothesis for the 7 participants placed randomly 1:1 in the jawline injection arm was that there would be no statistically significant change in the unblinded physician Jawline Rating Scale Assessment at baseline versus four weeks after last injection; Test type: Superiority; p = 0.00000031, t-test, 2 sided — The threshold for statistical significance was p = 0.05; The df = 13 for arm 1 (jawline injections) analysis of Jawline Rating Scale Assessments given by unblinded physician; Mean Difference (Final Values) = -1.0, Standard Deviation 0.497 — Treatment Difference = 4 Weeks after last injection - Baseline
Statistical Analysis 2: Comparison: Both Jawline and Lateral (Zygomatic) Cheek Area Injections; The null hypothesis for the 7 participants placed randomly 1:1 in the jawline and lateral (zygomatic) cheek area injections arm was that there would be no statistically significant change in the unblinded physician Jawline Rating Scale Assessment at baseline versus four weeks after last injection; Test type: Superiority; p = 0.0000728, t-test, 2 sided — The threshold for statistical significance was p = 0.05; The df = 13 for jawline and lateral (zygomatic) cheek area injections arm analysis of Jawline Rating Scale Assessments given by unblinded physician; Mean Difference (Final Values) = -0.714, Standard Deviation 0.497 — Treatment Difference = 4 Weeks after last injection - Baseline

3. Secondary Outcome: Subject Jawline Rating Scale (JRS) Assessment on Scale of 0 to 4 at Baseline Versus 4 Weeks After Last Injection.
Description: One of the secondary outcomes is a reduction of 1 or more points of the Jawline Rating Scale (JRS) Assessment (on a scale of 0 to 4) at baseline versus that at 4 weeks from the last injection (whether initial or touch-up) based on each subjects' ratings. (A lower number will mean a better outcome) To clarify the Time Point "4 Weeks from last injection" it means 8 to 12 weeks after baseline as subjects were eligible for treatment 4 weeks after baseline and possible retreatment 8 weeks after baseline. The study wanted to capture results 4 weeks after last injection.
  Scale Range Description 0 = No sagging
  1. = Mild sagging
  2. = Moderate sagging
  3. = Severe sagging
  4. = Very Severe sagging
Time Frame: Baseline to 4 weeks after last injection.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Jawline Injections | Both Jawline and Lateral (Zygomatic) Cheek Area Injections
Number analyzed (Participants) | 7 | 7
score on a scale
  Mean Jawling Rating Scores at Baseline | 2.286 (0.469) | 2.429 (0.514)
  Mean Jawline Rating Scores at 4 weeks after last injection | 1.714 (0.611) | 1.714 (0.726)
  Mean Reduction in Jawline Rating Score Baseline vs 4 Weeks after last injection | .571 (.545) | .714 (.629)
Statistical Analysis 1: Comparison: Jawline Injections; The null hypothesis for the 7 participants placed randomly 1:1 in the jawline injection arm was that there would be no statistically significant change in the subjects' Jawline Rating Scale Assessment at baseline versus four weeks after last injection; Test type: Superiority; p = 0.014, t-test, 2 sided — The threshold for statistical significance was p = 0.05; The df = 13 for jawline injections analysis of Jawline Rating Scale Assessments given by subjects; Mean Difference (Final Values) = -0.571, Standard Deviation 0.611 — Treatment Difference = 4 Weeks after last injection - Baseline
Statistical Analysis 2: Comparison: Both Jawline and Lateral (Zygomatic) Cheek Area Injections; The null hypothesis for the 7 participants placed randomly 1:1 in the jawline and lateral (zygomatic) cheek area injections arm was that there would be no statistically significant change in the subjects' Jawline Rating Scale Assessment at baseline versus four weeks after last injection; Test type: Superiority; p = 0.0065, t-test, 2 sided — The threshold for statistical significance was p = 0.05; The df = 13 for jawline and lateral (zygomatic) cheek area injections analysis of Jawline Rating Scale Assessments given by the subjects; Mean Difference (Final Values) = -0.714, Standard Deviation 0.726 — Treatment Difference = 4 Weeks after last injection - Baseline

4. Secondary Outcome: Number of Participants With Abnormal Confrontational Visual Fields Exam Findings
Description: -Ophthalmologic exams that include Confrontational Visual Fields Exam will be performed prior to any treatment, 30 minutes after treatment, and at all follow up in-person visits.
Time Frame: From initial treatment visit until12 weeks post last injection
Measure: Count of Participants; unit: Participants
Arm/Group | Jawline Injections | Both Jawline and Lateral (Zygomatic) Cheek Area Injections
Number analyzed (Participants) | 7 | 7
Participants | 0 | 0

5. Secondary Outcome: Number of Participants With Abnormal Eye Exam Findings
Description: -Ophthalmologic exams that include Snellen Eye Exam will be performed prior to any treatment, 30 minutes after treatment, and at all follow up in-person visits. The Snellen Eye Exam measures visual acuity, by reading a Snellen chart from 20 feet away. The farther down the chart the patient can read, the better their visual acuity is.
Time Frame: From initial treatment visit until12 weeks post last injection
Measure: Count of Participants; unit: Participants
Arm/Group | Jawline Injections | Both Jawline and Lateral (Zygomatic) Cheek Area Injections
Number analyzed (Participants) | 7 | 7
Participants | 0 | 0

6. Secondary Outcome: Number of Participants With Abnormal Ocular Motility Exam Findings
Description: -Ophthalmologic exams that include Ocular Motility Exam will be performed prior to any treatment, 30 minutes after treatment, and at all follow up in-person visits. Ocular motility examination is a binocular exam without the patient's glasses. Each eye of the subject is assessed for abnormalities in six positions of gaze: elevation upper lateral, elevation upper medial, elevation central, depression inferior lateral, depression inferior medial, and depression central.
Time Frame: From initial treatment visit until 12 weeks post final injection
Measure: Count of Participants; unit: Participants
Arm/Group | Jawline Injections | Both Jawline and Lateral (Zygomatic) Cheek Area Injections
Number analyzed (Participants) | 7 | 7
Participants | 0 | 0

7. Secondary Outcome: Number of Participants With Abnormal Cranial Nerves II, III, IV and VII Assessments Findings
Description: To further assess vision and oculomotor function, cranial nerves II, III, IV, and VII will be assessed (left and right sides separately). To assess lower face function, cranial nerves V, VII, IX, X and XII will be assessed. Individual tests will be rated (normal, abnormal that is not clinically significant, and abnormal that is clinically significant) assessing the function of the cranial nerves. These exams will be performed prior to any treatment, 30 minutes after treatment, and at all follow up visits.
Time Frame: From initial treatment visit until 12 weeks post last injection
Measure: Number; unit: participants
Arm/Group | Jawline Injections | Both Jawline and Lateral (Zygomatic) Cheek Area Injections
Number analyzed (Participants) | 7 | 7
participants | 1 | 0

8. Secondary Outcome: Number of Participants With Adverse Events
Description: Adverse events will be recorded until 12 months after last treatment. All study visits will assess Adverse Events: Treatment visits, 72 hr post Treatments, Week 2, Week 4, Week 8, Week 12/16, 6 Month and 12 Month follow-up visits.
Time Frame: From initial treatment visit until 12 months after last injection treatment
Measure: Number; unit: number of subjects with Adverse Events
Arm/Group | Jawline Injections | Both Jawline and Lateral (Zygomatic) Cheek Area Injections
Number analyzed (Participants) | 7 | 7
number of subjects with Adverse Events
  Mild Bruising | 2 | 6
  Mild Discomfort With Chewing | 6 | 3
  Mild Jaw Ache | 4 | 5
  Moderate Jaw Ache | 1 | 0
  Moderate Discomfort With Chewing | 1 | 0
  Swelling | 0 | 2
  Lumps/Bumps | 1 | 2
  Redness | 0 | 1
  Firmness | 2 | 3
  Headache | 1 | 0
  Cheek Pain | 0 | 3
  Ear Ache | 1 | 0
  Inability to Fully Extend Jaw | 1 | 0
  Bilateral Eyelid Drooping | 0 | 1
  Basal Cell Carcinoma | 0 | 2
  Right Arm and Right Leg Numbness | 0 | 1
  Moderate Bruising | 0 | 1

9. Secondary Outcome: Blinded Physician Jawline Rating Scale (JRS) Assessment on Scale of 0 to 4 for Group 1 (Jawline Injections) Versus Group 2 (Jawline and Lateral Zygomatic Cheek Area Injections) at 4 Weeks After Last Injection.
Description: One of the secondary outcomes is a statistically significant difference of the Jawline Rating Scale (JRS) Assessment (on a scale of 0 to 4) when comparing group 1 (Jawline Injections) and group 2 (Jawline and Lateral Zygomatic Cheek Area Injections) 4 weeks from the last injection (whether initial or touch-up) based on one blinded dermatologist rating. (A lower number will mean a better outcome). Photos will be taken at Baseline and 4 weeks after last injection treatment
Time Frame: From Baseline to 4 weeks after last injection
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Jawline Injections | Both Jawline and Lateral (Zygomatic) Cheek Area Injections
Number analyzed (Participants) | 7 | 7
score on a scale | 1.857 (.8644) | 1.857 (.8644)

10. Secondary Outcome: Unblinded Physician Jawline Rating Scale (JRS) Assessment on Scale of 0 to 4 for Group 1 (Jawline Injections) Versus Group 2 (Jawline and Lateral Zygomatic Cheek Area Injections) at 4 Weeks After Last Injection.
Description: One of the secondary outcomes is a statistically significant difference of the Jawline Rating Scale (JRS) Assessment (on a scale of 0 to 4) when comparing group 1 (Jawline Injections) and group 2 (Jawline and Lateral Zygomatic Cheek Area Injections) 4 weeks from the last injection (whether initial or touch-up) based on one unblinded dermatologist rating. (A lower number will mean a better outcome)
Time Frame: From Baseline until 4 weeks after last injection
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Jawline Injections | Both Jawline and Lateral (Zygomatic) Cheek Area Injections
Number analyzed (Participants) | 7 | 7
score on a scale | 1.357 (.497) | 1.643 (.497)

11. Secondary Outcome: Subject Jawline Rating Scale (JRS) Assessment on Scale of 0 to 4 for Group 1 (Jawline Injections) Versus Group 2 (Jawline and Lateral Zygomatic Cheek Area Injections) at 4 Weeks After Last Injection.
Description: One of the secondary outcomes is a statistically significant difference of the Jawline Rating Scale (JRS) Assessment (on a scale of 0 to 4) when comparing group 1 (Jawline Injections) and group 2 (Jawline and Lateral Zygomatic Cheek Area Injections) 4 weeks from the last injection (whether initial or touch-up) based on subjects' ratings. (A lower number will mean a better outcome)
Time Frame: From Baseline until 4 weeks after last injection
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Jawline Injections | Both Jawline and Lateral (Zygomatic) Cheek Area Injections
Number analyzed (Participants) | 7 | 7
score on a scale | 1.714 (.611) | 1.714 (.726)

ADVERSE EVENTS:
Time Frame: 12 months after last treatment
Description: Adverse events were monitored at every patient visit and through patient safety diaries completed daily for 1 month following treatment.
Arm/Group | Jawline Injections | Both Jawline and Lateral (Zygomatic) Cheek Area Injections
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 7/7 | 7/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Jawline Injections (N=7) | Both Jawline and Lateral (Zygomatic) Cheek Area Injections (N=7)
Mild bruising (Skin and subcutaneous tissue disorders) | 2 (2) | 6 (9)
mild discomfort with chewing (Skin and subcutaneous tissue disorders) | 6 (6) | 3 (3)
Mild jaw ache (Skin and subcutaneous tissue disorders) | 4 (5) | 5 (5)
Moderate jaw ache (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Moderate discomfort with chewing (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Swelling (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Lumps/bumps mass or nodule (Skin and subcutaneous tissue disorders) | 1 (2) | 2 (2)
Redness (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Firmness (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3)
Headache (Nervous system disorders) | 1 (2) | 0 (0)
Cheek pain (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
Ear ache (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Inability to fully extend jaw (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Bilateral eyelid droop (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Basal Cell Carcinoma (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Moderate bruising (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
arm or leg numbness (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The limitations and caveats are the following: Small sample size, limited to females only, interrupted by COVID with some discontinuous visits, 2 patients were evaluated as mild at baseline by the blinded physician and they should have been excluded.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-04-24): https://cdn.clinicaltrials.gov/large-docs/66/NCT04389866/Prot_SAP_000.pdf
  • Informed Consent Form (2020-07-20): https://cdn.clinicaltrials.gov/large-docs/66/NCT04389866/ICF_001.pdf